CLINICAL TRIAL: NCT01587313
Title: A Four-arm, Single Dose, Two-Period, Pharmacokinetic Study of BiDil SR and IR Capsules and Commercial BiDil Tablets
Brief Title: A Comparison of Various Combinations of BiDil Capsules and BiDil Tablets in Healthy Human Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arbor Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: AR06.004
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: hydralazine; isosorbide; bidil; volunteers; pharmacokinetic profile
MeSH Terms: interventions — Isosorbide Dinitrate; Hydralazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): ISDN/HYD 2 SR caps crossover to 1 IR cap at 8 am
  Interventions: Drug: Isosorbide dinitrate / hydralazine capsules
- Group 2 (Experimental): ISDN/HYD 2 SR caps crossover to 1 IR cap at 5 pm
  Interventions: Drug: Isosorbide dinitrate / hydralazine capsules
- Group 3 (Experimental): ISDN/HYD 2 SR caps crossover to 1 IR cap at 8 pm
  Interventions: Drug: Isosorbide dinitrate / hydralazine capsules
- Group 4 (Active Comparator): ISDN/HYD 1 IR cap and two SR caps at 8 am crossover to Day 8: BiDil Tablet tid
  Interventions: Drug: Isosorbide dinitrate / hydralazine capsules

INTERVENTIONS:
Drug: Isosorbide dinitrate / hydralazine capsules — Group 1: Day 1:Two SR capsules; Day 8: One IR capsule Group 2: Day 1:Two SR capsules; Day 8: One IR capsule Group 3: Day 1:Two SR capsules; Day 8: One IR capsule Group 4: Day 1:One IR capsule and two SR capsules; Day 8: Commercial BiDil Tablet tid
  Other Names: BiDil tablets; ISDN/HYD

SUMMARY:
This is a single center, open-label, two-period study. There will be nine healthy human volunteers arbitrarily assigned to one of four groups. The study objective is to compare the action of various combinations of BiDil extended-release capsules and commercial BiDil Tablets in the body over a period of time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, nonsmoking, slow acetylator (as determined by caffeine metabolite assay) males or females between the ages of 18 to 40 years inclusive.
* Body weight at least 150 pounds and Body Mass Index between 18.5 and 30 kg/m2.
* Medical history, physical examination, and clinical laboratory test results indicating either normal vital organ/endocrine functions, or no clinically significant abnormalities.
* Clinical laboratory testing negative for: HIV, Hepatitis B surface antigen and Hepatitis C antibody.
* Urine testing negative for drugs of abuse (including, but not limited to marijuana, amphetamines, barbiturates and cocaine).
* Negative urine cotinine test and negative saliva alcohol test.
* Negative urine HCG test, consistent with no pregnancy (females only).
* For female subjects, a recent history of menses that is regular for the individual (24 36 day cycles).
* Females participating in this study must be:
* unable to have children (e.g., post-menopausal, tubal ligation, hysterectomy) OR
* willing to remain abstinent [not engage in sexual intercourse for the duration of the screening period and throughout the study, and for 14 days after the last dose] OR
* willing to use two effective barrier methods of birth control (partner using condom and female using IUD, diaphragm plus spermicide, or contraceptive sponge).
* Ability to grant voluntary informed consent to participate in the study.

Exclusion Criteria:

* Known history or presence of any clinically significant medical condition.
* Known or suspected carcinoma.
* Use of prescription or OTC drug(s), other than acetaminophen, within two weeks of first dose of study drug and throughout study unless approved by the investigator or sponsor.
* Use of alcohol or caffeine containing products within 48 hours of each dose of study drug.
* History of, or evidence of clinically significant medical condition, including, but not limited to hepatic, renal, cardiac, vascular, gastrointestinal, or thyroid disease, diabetes, epilepsy, respiratory or hematological disease, acute narrow angle glaucoma or psychiatric disorder which, in the opinion of the Investigator would confound the study results or present a risk to the subject.
* History of alcohol or drug abuse within one year of study participation.
* Presence of, or known hypersensitivity, allergy, idiosyncratic reaction or adverse reaction to caffeine, ISDN, hydralazine HCl, or any compounds with similar chemical characteristics.
* Received an investigational drug within 30 days of the first dose in this study.
* Blood pressure less than 110/70 mm Hg at screening or at Day 1 prior to dosing.
* Donated one pint or more of blood or donated platelets within 30 days of the first dose in this study.
* Any subject who, in the opinion of the Investigator, cannot follow instructions.
* With regard to females; pregnancy, lactation, or the use of hormonal contraception.
* History of lupus erythematous or lupus like syndrome.
* Use of herbal preparations or use of phosphodiesterase inhibitors.
* Employee of the Sponsor or CRO.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Area under the plasma/blood concentration versus time curve, as calculated by the linear trapezoidal method for Hydralazine and ISDN and metabolites. | from time zero (0) to 24 hr

CONTACTS AND LOCATIONS:
Overall Officials: Gregory J Tracey, MD, Principal Investigator — Frontage Laboratories, Inc.
Locations (1):
- Frontage Cinical Services, Hackensack, New Jersey, United States